CLINICAL TRIAL: NCT02426359
Title: Safety and Efficacy Study of Q301 in Moderate to Severe Atopic Dermatitis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qurient Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Q301-ADP2-US-01
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-05

CONDITIONS: Moderate to Severe Atopic Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Q301 Cream (Experimental): Q301 Cream
  Interventions: Drug: Q301 Cream
- Vehicle (Placebo Comparator): Vehicle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Q301 Cream
  Arms: Q301 Cream
Drug: Placebo
  Arms: Vehicle

SUMMARY:
This is a randomized, double-blind, vehicle-controlled, parallel-group comparison study to evaluate the safety and efficacy of Q301 Cream vs. vehicle in adult subjects with moderate to severe AD. Study drug (Q301 Cream or vehicle) will be administered topically twice a day for 8 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 or older
2. Subjects with a clinical diagnosis of AD according to the Hanifin and Rajka Criteria by a board certified/eligible dermatologist
3. Subjects with IGA score 3 or 4 corresponding to moderate to severe AD at screening and baseline visits

Exclusion Criteria:

1. Subjects who had topical treatment with corticosteroids within 1 week before randomization
2. Subjects who had systemic treatment with corticosteroids or cyclosporine or other immunosuppressive treatment within 4 weeks before randomization
3. Subjects who had ultraviolet irradiation (including photopheresis) within 4 weeks before screening
4. Subjects who participated in another drug trial within 4 weeks before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who have the IGA score of 0 or 1 | Week 8

SECONDARY OUTCOMES:
Percent change from baseline on the VAS for pruritus | Week 8
Percent change from baseline on the EASI | Week 8
Percent change from baseline on the SCORAD | Week 8
Percent change from baseline on the DLQI | Week 8

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Denver, Colorado
  - Berlin, New Jersey
  - East Windsor, New Jersey
  - Buffalo, New York
  - Winston-Salem, North Carolina
  - Austin, Texas
  - College Station, Texas